CLINICAL TRIAL: NCT05986305
Title: Improving the Health of Parents and Their Adolescent and Transition-age Youth With Intellectual and Developmental Disabilities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0739
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Go Act (Active Comparator): Go Act is structured as a small group intervention for parents, consisting of four 60-minute sessions occurring over a 4-week period.
  Interventions: Behavioral: Go Act
- Peer (Active Comparator): Peer is structured as a small group intervention for parents, consisting of four 60-minute sessions occurring over a 4-week period.
  Interventions: Behavioral: Peer

INTERVENTIONS:
Behavioral: Go Act — Go Act sessions address becoming a parent who can 'Go Act,' caring for one's self as a parent, understanding and managing youth health needs, working with health providers as partners, and working with other service providers such as schools and vocational services. The intervention uses motivational interviewing, story-telling with self-disclosure, psycho-education introduced with a know-want to know-learned strategy, problem-solving, role play, and practice outside of class.
  Arms: Go Act
Behavioral: Peer — During Peer sessions facilitators lay ground rules for respectful and confidential sharing and encourage group discussion. The group provides a format to make personal connections through shared identity. Participants may discuss strategies for individualized advocacy, so that they learn from the experiences of others.
  Arms: Peer

SUMMARY:
This study will determine the comparative effectiveness of Go Act, a tailored advocacy curriculum versus Peer parent-directed peer learning for increasing parent activation for parents of youth with intellectual and developmental disabilities. Second, it will determine the comparative effectiveness of the two study arms for improving parent and youth health outcomes while assessing whether parent activation serves as a mechanism that mediates their effects on health outcomes.

DETAILED DESCRIPTION:
A well-functioning system of care should provide a broad array of services that can support families with a child with complex health care needs. Nonetheless, adolescents and transition age youth with intellectual and developmental disabilities experience rates of unmet need for health care up to 6 times higher than others resulting in poor health and quality of life for themselves and their families.

The system of care approach has achieved positive impacts for children with intellectual and developmental disabilities and their families, but updates call for training to help parents develop advocacy skills on behalf of their children. Prior research on diverse populations indicates that parent advocacy skills are a promising target for increasing parent self-efficacy, which in turn is associated with better parent and youth health outcomes. Parent advocacy skills can be increased through a psycho-educational advocacy skills curriculum or through parent-directed peer-learning. However, the comparative effectiveness of these two strategies for families raising youth with intellectual and developmental disabilities is not yet known.

This study has two objectives. First, it will determine the comparative effectiveness of Go Act, a tailored advocacy curriculum versus Peer parent-directed peer learning for increasing parent activation for parents of youth with intellectual and developmental disabilities . Second, it will determine the comparative effectiveness of the two study arms for improving parent and youth health outcomes while assessing whether parent activation serves as a mechanism that mediates their effects on health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Parents

* Raising an adolescent or young adult child (age 11-27), with diagnosed or suspected intellectual or developmental disability
* Able to attend group sessions
* Able to give informed consent
* Resident of any state except New York or Illinois due to electronic signature law

Youth

* Being between the ages of 11 and 27
* Having diagnosed or suspected intellectual or developmental disability

Exclusion Criteria:

Parents

• Having evidence of emergency mental health needs

Ages: 11 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 406 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change in parent activation | up to18 months after intervention
  The Parent Patient Activation Measure will be used to capture parent activation on behalf of their child (mean score=70) at 6, 12 and 18 months after intervention. The Parent Patient Activation Measure is a parent self-report 13-item scale with 4-level likert responses and scores ranging from 0 to 100.
Difference in change in youth social functioning- life satisfaction | up to18 months after intervention
  Youth social functioning will be assessed using the NIH Patient-Reported Outcomes Measurement Information System for children life satisfaction measure at 6, 12 and 18 months after intervention.
Difference in change in parent depression | up to 18 months after intervention
  Parent depression will be measured with the 8-item Patient Health Questionnaire at 6, 12 and 18 months after intervention. The Patient Health Questionnaire is scored from 0 to 24.

SECONDARY OUTCOMES:
Difference in change in parenting self-efficacy | up to 18 months after intervention
  The Tool to Measure Parenting Self-Efficacy will be used to assess parent self-efficacy at 6, 12 and 18 months after intervention. The Tool to Measure Parenting Self-Efficacy short version consists of 36-items rated on an 11-point likert scale, from 0 to 10 completely disagree to completely agree. Individual items are summed to create a total score, with higher scores indicating greater feelings of parenting self-efficacy.
Difference in change in shared decision-making | up to 18 months after intervention
  Shared decision-making will be assessed using a three-item scale from the National Survey of Children's Health at 6, 12 and 18 months after intervention. Respondents report on a 4-point likert scale (never, sometimes, usually, or always) whether they feel that they 1) discuss with providers a range of treatment options; 2) are encouraged to raise concerns; 3) make treatment choices together. Mean scores range from 1 to 4 never to always.
Difference in change in alliance | up to 18 months after intervention
  The adapted Parenting Alliance Inventory will be used to measure parent-teacher alliance at 6, 12 and 18 months after intervention. The Parenting Alliance Inventory was adapted to focus on parent-teacher alliance, and consists of 20 items scored on a 5-point likert scale, producing a mean score between 1 and 5 never to always.
Difference in change in goal attainment | up to 18 months after intervention
  Goal attainment will be assessed with the psychometric equivalence tested goal attainment scale at 6, 12 and 18 months after intervention. The goal attainment scale measurement system is based on a 5-point response scale ranging from -2 (worse expected outcome) to 2 (best expected outcome).
Difference in change in stress | up to 18 months after intervention
  Parent stress will be measured with the 17-item Parental Stress Scale at 6, 12 and 18 months after intervention. Mean scores range from 1 to 5 with higher scores indicating higher stress.
Difference in change in observed parent activation | up to18 months after intervention
  Observed parent activation will be assessed through audio-recorded parent-physician conversations at 6, 12 and 18 months after intervention. Evidence of parent activation will be examined: 1) providing context, 2) giving feedback, and 3) asking questions. Audio-recordings will be transcribed and a coding manual created.
Difference in change in youth social functioning- meaning & purpose | up to 18 months after intervention
  Youth social functioning will additionally be assessed using the NIH Patient-Reported Outcomes Measurement Information System for children meaning and purpose measure at 6, 12 and 18 months after intervention.
Difference in change in youth unmet need for care | up to 18 months after intervention
  Unmet need for care will be assessed using a three-item scale from the National Survey of Children's Health items at 6, 12 and 18 months after intervention. Respondents report 1) that they needed but did not receive care (yes/no), 2) types of care not received, and 3) reasons for not receiving care. Counts of reasons (0 to 6) are summed for each of 5 types of care.
Difference in change in youth psychiatric crisis care use | up to 18 months after intervention
  Psychiatric crisis care use will be measured by number of emergency department visits at 6, 12 and 18 months after intervention.
Difference in change in number of inpatient psychiatric stays | up to 18 months after intervention
  Inpatient psychiatric stays will be measured by number of stays at 6, 12 and 18 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen C Thomas, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - The Carolina Institute for Developmental Disabilities, Carrboro, North Carolina
  - UNC Adult Psychiatry Clinic, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board, Independent Ethics Committee, or Research Ethics Board, as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: ICF
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved Institutional Review Board, Independent Ethics Committee, or Research Ethics Board and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.